CLINICAL TRIAL: NCT06192992
Title: Regional Blood Flow During Peripheral Heating
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jeffrey Moore, Adjunct Professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: PHTBloodFlow
Record Dates: First submitted 2022-05-31; First posted 2024-01-05 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Blood Flow
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (Sham Comparator): Blood flow without heating
  Interventions: Other: Sham
- Two feet (Experimental): Blood flow during heating of two feet
  Interventions: Other: Peripheral heating of 2 feet

INTERVENTIONS:
Other: Peripheral heating of 2 feet — Heating of both feet
  Arms: Two feet
Other: Sham — No heating
  Arms: Sham

SUMMARY:
Blood flow through the popliteal, brachial, and carotid arteries during peripheral heating of the feet

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years

Exclusion Criteria:

* open wounds on feet or legs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Blood flow through the popliteal, brachial, and carotid arteries | 30 minute
  blood flow through arteries measured via ultrasound doppler (mL/s)

CONTACTS AND LOCATIONS:
Locations (1):
- Jeff Moore, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No